CLINICAL TRIAL: NCT06556056
Title: Exploratory, Prospective, Three-arm, Interventional, Comparative, Randomized, Double-blind, Placebo-controlled, Safety, Efficacy and In-use Tolerability Study of Hair Growth Product(s) in Patients With Mild to Moderate Androgenic Alopecia: (Grade I to III)
Brief Title: An Exploratory Clinical Study to Assess Safety, Efficacy and In-Use Tolerability of Three Different Hair Growth Products in Patients With Mild to Moderate Androgenic Alopecia (Grade I to III)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Zywie Ventures Privated Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NB240029-ZV
Record Dates: First submitted 2024-08-02; First posted 2024-08-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-08

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SesZen-Bio Serum (Experimental): Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Dosage form: liquid Frequency: Daily Night application. Rout of administration: Topical
  Interventions: Other: SesZen-Bio Serum
- Minoxidil Hair Serum (1%) (Active Comparator): Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Dosage form: Liquid Frequency: Daily Night Application Rout of administration: Topical
  Interventions: Other: Minoxidil hair serum (1%)
- Placebo (Placebo Comparator): Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Dosage form: Liquid Frequency: Daily Night Application Rout of administration: Topical
  Interventions: Other: Placebo
- Liposomal Form of SesZenBio (Experimental): Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Frequency: Daily Night Application Rout of administration: Topical
  Interventions: Other: Liposomal Form of SesZenBio
- Minoxidil Hair Serum (5%) (Experimental): Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Frequency: Daily Night Application Rout of administration: Topical
  Interventions: Other: Minoxidil Hair Serum (5%)
- SesZen-Bio Serum + SesZen-Bio 350 mg extract (Experimental): Mode of Usage of serum: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Frequency: Daily Night Application Rout of administration: Topical Mode of Usage of Capsule: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Frequency: One time daily after meal Rout of administration: Oral
  Interventions: Other: SesZen-Bio Serum + SesZen-Bio 350 mg extract

INTERVENTIONS:
Other: SesZen-Bio Serum — Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Dosage form: Liduid Frequency: Daily Night application. Route of administration: Topical
  Arms: SesZen-Bio Serum
Other: Minoxidil hair serum (1%) — Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Dosage form: Liquid Frequency: Daily Night Application Route of administration: Topical
  Arms: Minoxidil Hair Serum (1%)
Other: Placebo — Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Dosage form: Liquid Frequency: Daily Night Application Route of administration: Topical
  Arms: Placebo
Other: Liposomal Form of SesZenBio — Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Frequency: Daily Night Application Rout of administration: Topical
  Arms: Liposomal Form of SesZenBio
Other: Minoxidil Hair Serum (5%) — Mode of Usage: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Frequency: Daily Night Application Rout of administration: Topical
  Arms: Minoxidil Hair Serum (5%)
Other: SesZen-Bio Serum + SesZen-Bio 350 mg extract — Mode of Usage of serum: Dispense a small amount of serum directly onto your fingertips and gently massage it into the roots and scalp using circular motions to ensure even distribution and absorption. Continue this process across your entire scalp, focusing on areas that need the most attention. Avoid rinsing the serum out; instead, allow it to absorb fully.
  Frequency: Daily Night Application Rout of administration: Topical Mode of Usage of Capsule: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Frequency: One time daily after meal Rout of administration: Oral
  Arms: SesZen-Bio Serum + SesZen-Bio 350 mg extract

SUMMARY:
This is an exploratory, prospective, three-arm, interventional, comparative, randomized, double-blind, placebo-controlled, safety, efficacy and in-use tolerability study of hair growth products in the patients mild to moderate androgenic alopecia (Grade I to III).

DETAILED DESCRIPTION:
A total of up to 54 patients (18 patients/arm) preferably equal number of male and female will be enrolled to ensure a total of 45 patients (15 patients/ arm) to complete the study. Additional arm 4, 18subjects was added to complete 15, as an open-label, exploratory, prospective, interventional arm to evaluate the efficacy and safety of the liposomal form of SesZen Bio serum, with comparative reference to the Minoxidil arm. Following further, two more open-label arms-Arm 5 and Arm 6- have now been incorporated into the study to evaluate the comparative efficacy and safety of 5% Minoxidil and combination therapy consisting of SesZen Bio capsules (350 mg standardized extract) with the SesZen Bio serum. Each arm will enrol 18 healthy subjects to achieve 15 evaluable subjects per arm

There will be total of 8 visits during the study. The duration of the study will be 180 days (6 months) from the enrolment.

visit 1(Day -04): Screening, Tattoo creation, hair growth measurement. Visit 02(Day 01): Enrolment, hair growth rate measurement, hair length, hair thickness, hair density, scalp condition for keratin measurement, A: T ratio, number of new hairs, number of hair fall from root, hair root strength, general appearance of hair, general appearance of scalp, earlier product perception questionnaire, global pictures of head crown.

Visit 03 (Day 45): Hair Length, hair thickness, hair density, scalp condition for keratin measurement, hair regrowth, number of hair fall from root, number of new hairs from the full scalp, AG affected, hair root strength, general appearance of hair, general appearance of scalp, product perception questionnaire, global pictures of head crown.

Visit 04 (Day 87): Tattoo creation, hair growth measurement Visit 05 [Day 90 (03 days from visit 04)]:Hair growth rate measurement, hair length, hair thickness, hair density, scalp condition for keratin measurement, A: T ratio, hair regrowth, number of new hairs, number of hair fall from root, hair root strength, general appearance of hair, general appearance of scalp, product perception questionnaire, digital photographs of global pictures head crown.

Visit 06 (Day 135): Hair length, hair thickness, hair density, scalp condition for keratin measurement, hair regrowth, number of hair fall from root, number of new hair, hair root strength from root, general appearance of hair, general appearance of scalp, product perception questionnaire, digital photographs of global pictures head crown.

Visit 07 (Day 177) : Tattoo creation, hair growth measurement Visit 08: [Day 180 (03 days from Visit 07)]: Hair growth rate measurement, hair length, hair thickness, hair density, scalp condition for keratin measurement, A: T Ratio, number of new hair, hair regrowth, number of hair fall from root, hair root strength, general appearance of hair, general appearance of scalp, product perception questionnaire, global pictures of head crown

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25 to 45 years and above (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Females of childbearing potential must have a self-reported negative urine pregnancy.
4. Subject is in good general health as determined by the Investigator on the basis of medical history.
5. Patients having mild to moderate androgenic alopecia (Grade I to III) during clinical study and grade will be evaluated by the dermatologist by using Norwood-Hamilton classification and Ludwig pattern scale for female.
6. Female with 40-50 counts and male with 25 -30 counts of hair fall at screening.
7. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
8. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
9. Patients are willing to give written informed consent and are willing to follow the study procedure.
10. Patients who commit not to use any other medicated/ prescription shampoos/hair care products (containing Minoxidil), any other hair growth products or hair colour or dye, other than the test products for the entire duration of the study.
11. Willing to use test products throughout the study period.
12. Subject is willing and able to follow and allow study staff to performed study test methods.
13. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
14. Subject must be able to understand and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Subject have history of severe hair fall due to any clinically significant problems like anaemia, thyroid problems.
2. Subject have history of any dermatological condition of the scalp other than hair loss and dandruff.
3. Subject have history of any prior hair growth procedures (e.g. hair transplant or laser).
4. Subject who had taken topical treatment of hair loss for at least 4 weeks.
5. Subject who had taken any systemic treatment for at least 3 months.
6. History of alcohol or drug addiction.
7. Subject having history or resent condition of irritated or visibly inflamed scalp or severe scalp disease.
8. Subject having history or present condition of an allergic response to any cosmetic products, any other condition which could warrant exclusion from the study.
9. Pregnant or breast feeding or planning to become pregnant during the study period.
10. History of chronic illness which may influence the cutaneous state.
11. Subject have participated any clinical research study related to hair care products.
12. Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in hair thickness by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180.
  To assess the effectiveness of the test products in terms of change in hair thickness.
Change in hair density by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180.
  To assess the effectiveness of the test products in terms of change in hair density
Change in hair growth rate using CASLite Nova (instrumental analysis) | 04 before Day 01, Day 01, Day 87, Day 90, Day 177 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair growth rate

SECONDARY OUTCOMES:
Change in keratin measurement from scalp by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180.
  To evaluate the effectiveness of test products in terms of change in keratin measurement from scalp from Androgenic Alopecia affected targeted area and normal scalp- tattoo area
Change in hair length by using CASLite Nova (instrumental analysis) and calibrated ruler | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair length from androgenic alopecia affected targeted area and standard area
Change in A:T ratio by hair pluck test | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in A:T ratio by dermatologist
Change hair fall from root test by 60 seconds hair combing test | 04 before Day 01, Day 87, Day 90, Day 177 and on Day 180
  To assess the effectiveness of the test products in terms of change hair fall by dermatologist
Change in number of new hairs by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in number of new hairs
Change in hair regrowth by using CASLite Nova (instrumental analysis) | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair regrowth from androgenic alopecia affected targeted area
Change in hair root strength | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45 , Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair root strength by dermatologist.
Change in general appearance of hair volume | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair volume in which score done as small, medium, full
Change in general appearance of hair plasticity | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair plasticity in which score done as waved and average
Change in general appearance of hair density | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair density in which score as thinned and dense
Change in general appearance of hair dryness | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair dryness in which score done as 1= none, and 4= Excessive
Change in general appearance of hair shininess | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair shininess in which score done as 1= poor average and 3=good
Change in general appearance of hair smoothness | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair smoothness in which score done as 1= poor, and 3= good
Change in general appearance of hair oiliness | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair oiliness in which score done as 1= none and 4=excessive
Change in general appearance of hair strength | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair strength in which score done as poor, average and good
Change in general appearance of scalp Itchiness | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp Itchiness in which score done as none, mild, moderate and excessive
Change in general appearance of scalp redness | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp redness in which score done as none, mild, moderate and excessive
Change in general appearance of scalp roughness | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp roughness in which score done as none, mild, moderate and excessive
Change in general appearance of scalp scaliness | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp scaliness in which score done as none, mild, moderate and excessive
Change in general appearance of scalp dryness | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp dryness in which score done as 1= none, and 4=excessive
Change in products perception questionnaire in which 5-point Likert scale as 1= not at all and 5= to large extent | Before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  10. To evaluate the effectiveness of the test products in terms of change in products perception questionnaire
Change in tensile strength of hairs by TESTRONIX tensile tester (instrumental analysis) | Baseline before usage of test product on Day 01 and after usage of test product on Day 180.
  To assess the effectiveness of the test products in terms of change in tensile strength of hairs

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Private Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No